CLINICAL TRIAL: NCT02324192
Title: Hand Ultrasonography: Clinical and Functional Correlation in Symptomatic Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Natalia de Oliva Spolidoro Paschoal, Dr, Federal University of São Paulo
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: FUSaoPaulo002
Record Dates: First submitted 2014-12-09; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthritis
Keywords: Ultrasonography; clinical; hand
MeSH Terms: conditions — Osteoarthritis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal ultrasonography (Other): Patients with normal ultrasonography findings
  Interventions: Other: Ultrasonography
- Inflammatory ultrasonography (Other): Patients with inflammatory ultrasonography findings
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — imaging findings

SUMMARY:
Objective: To evaluate the correlation / association between inflammatory ultrasonography findings and clinical /functional assessment in symptomatic hand OA interphalangeal joints (IP). To evaluate the intra and interobserver reproducibility of ultrasound findings.

Methods: It was conducted a prospective study in 60 symptomatic hand OA patients. They were assessed in six times (T0, T1, T4, T8, T12 and T48 weeks) by "blind" observers (clinical and ultrasonography). The intra and interobserver reproducibility analysis was performed in 25% of the sample. Differences were considered as statistically significant when p< 0.05.

DETAILED DESCRIPTION:
Introduction Osteoarthritis (OA) is the most prevalent joint disease actually , hand OA is one of the characteristic subtypes. The estimated prevalence is 26% in over 70 years women. Treatment and follow-up of this disease have received less attention when compared to cases involving the knee and hip, probably because such involvement does not present with functional limitations as those seen in large joints.

For diagnosis and follow-up of hand OA the conventional radiography is used, although this exam give us an insight into just two planes of articulation and does not allow a reliable approach of tendons, muscles and other periarticular structures.

The ultrasound (US) appears as an emerging technique. More sensitive techniques are required for disease progression evaluation). It is a very useful imaging method, capable of showing early and late inflammation-related injuries and structural damage and is considered a great test to follow-up rheumatic diseases patients. Safe, easy to perform, low cost, fast and able to evaluate various sites attacked in the same turn, can be used in monitoring and evaluation of therapeutic response in these patients.

Some authors suggest that the sonographic evaluation is better than that of plain radiography, does not involve radiation and allows the joint evaluation at various sites. However, ultrasound still has limited use in hand OA compared to this use in inflammatory joint diseases.

The objectives of this study were to evaluate the correlation / association between ultrasonographic findings of inflammatory synovial hypertrophy and power Doppler of the interphalangeal joints(IP) and clinical and functional variables in patients with hand OA and test the intra and interobserver reproducibility of these ultrasonographic findings

Material and methods. A prospective study of ultrasonography in 60 patients with hand OA of was performed.

The inclusion criteria were: diagnosis of hand OA, according to the criteria of the American College of Rheumatology (ACR) with involvement of proximal and / or distal IP joints; more than 40 years old; visual analog scale of pain (VAS of 0-10 cm) in the joint of study between 3-8cm; and agree and sign the Consent Term of the study.

Exclusion criteria were: changed the use of oral corticosteroids and nonsteroidal anti-inflammatory drugs in the last thirty days; changed the treatment of OA in the last two months (including drug and rehabilitation); radiography of hands suggesting interphalangeal arthropathy of other etiology (psoriatic arthritis, microcrystalline arthropathy).

The most symptomatic joint was evaluated 60 patients in the study. Patients were evaluated at six times, having been made, so 360 assessments. Each in its dorsal recess (360) and palmar (360) recesses, accounting 720 joint recesses at the end of the study. Patients were from the outpatient rheumatology clinic of the Federal University of São Paulo (UNIFESP), Paulista Medical School, São Paulo, Brazil. The study was approved by the Research Ethics Committee of this Institution.

Evaluation Two "blind" observers (a clinical and a ultrasonography) evaluated the most symptomatic IP joint in the first assessment at the following times: T0, T1, T4, T8, T12 and T48 weeks.

At time 0 (T0) evaluation demographic data were collected and a plain radiograph of the hands was performed in anteroposterior view.

Clinical Evaluation Patients were evaluated in the six times according to the following assessment tools: visual analogue scale(VAS) of pain at rest of the studied joint (VASr 0-10 cm); VAS of the joint on movement(VASm of 0-10cm); VAS of joint swelling according to the evaluator (VASs 0-10cm); joint goniometry; need for analgesics (paracetamol 750mg daily average expressed in tablets / day); handgrip strength by Jamar dynamometer grip (instruction manual, PC 5030J1- Preston / Trenton, Ontario Canada; Mathiowetz, 1984) involving the studied joint hand; pinch strength (pulp-pulp, tripod and key) through the dynamometer Pinch Gauge (instruction manual, A853-4-Smith & Nephew / Germantown, United States of America; Mathiowetz, 1984) in the studied finger; hand function assessed by the Brazilian version of two functional questionnaires, the COCHIN questionnaire and AUSCAN Index.

Ultrasound evaluation

The ultrasonography evaluation was performed after each clinical assessment, on all six times of evaluation by an experienced sonographer in musculoskeletal US. The US examination was carried out using a MyLab 60 Xvision (Esaote, Biomedica - Genova, Italy) using a linear transducer frequency 10-18 megahertz(MHz). The following ultrasonography parameters were evaluated: Synovial Hypertrophy (SH):

Quantitative measurement of synovial hypertrophy(SH): This measurement was made between the bone surface to the the joint capsule of the dorsal and palmar recess in each assessment and expressed in millimeters (mm).

Semiquantitative measurement of SH: assessed by a semiquantitative score ranging from 0 to 3, modified for the proximal IP (PIP) and distal (IFD) from the score created by Szkudlarek and collaborators in 2003. According to this score:Grade 0 = no fluid; B, grade 1 = minimal amount of fluid; C, grade 2 = moderate amount of fluid (without distension of the joint capsule); D, grade 3 = extensive amount of fluid (with distension of the joint capsule). Scores 0 or 1 were considered normaland pathological scores 2 or 3.

Synovial Blood Flow: estimated by the presence of signal power Doppler (PD) which was also graded 0-3. Grade 0 = no flow in the synovium; grade 1 = single vessel signals; grade 2 = confluent vessel signals in less than half of the area of the synovium; grade 3 = vessel signals in more than half of the area of the synovium. The pulse repetition frequency (PRF) was maintained between 500 and 1000 Hz The frequency varied between 6.3 and 10 MHz. It was considered normal grade 0 and pathological grade 1, 2 and 3.

Intraobserver and interobserver reproducibility of ultrasound evaluation Assessment of intra- and interobserver reproducibility was performed for quantitative and semiquantitative measures of SH and PD. This evaluation was done in 25% of the sample (90 joint recesses).

In this analysis two ultrasonographers were involved. The first was responsible for ultrasonographic evaluation of the entire sample. In addition, he was also responsible for conducting a second ultrasound measure used to assess intraobserver reproducibility. The second ultrasonographer was responsible for ultrasonographic evaluation used to assess inter-observer reproducibility. During the evaluation of the first ultrasonographer images were evaluated and then recorded. Such images recorded were identified with numbers (and not with the patient's name) and evaluated by the same ultrasonographer (first ultrasonographer) with more than 60 days interval. The second ultrasonographer did the ultrasound evaluation in images recorded by the first ultrasonographer completely independently.

Statistical Analysis Continuous data sample were described by mean and standard deviation (SD). Categorical data were expressed as frequencies and percentages. Continuous variables sample were tested with normality Kolmogorov-Smirnov test; Spearman correlation were used for continuous variables; Mann-Whitney test for the association between continuous and categorical variables and the chi-square test for categorical variables.

Reproducibility assessment for ultrasonography measurements was performed using the kappa test and the intraclass correlation coefficient (ICC).

Differences were considered as statistically significant when p< 0.05

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hand OA, according to the criteria of the American College of Rheumatology (ACR) (Altman et al., 1990) with involvement of proximal and / or distal IP joints
* More than 40 years old
* Visual analog scale of pain (VAS of 0-10 cm) in the joint of study between 3-8cm
* And agree and sign the Consent Term of the study.

Exclusion Criteria:

* Changed the use of oral corticosteroids and nonsteroidal anti-inflammatory drugs in the last thirty days
* Changed the treatment of OA in the last two months (including drug and rehabilitation)
* Radiography of hands suggesting interphalangeal arthropathy of other etiology (psoriatic arthritis, microcrystalline arthropathy).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline - Correlation between VASr(Visual Analogic Scale of pain at rest 0-10cm) and ultrasonography findings(Grey Scale and power Doppler) at 1year in six times | 0,1,4,8,12 and 48 weeks

SECONDARY OUTCOMES:
Change from baseline - Correlation between VASs(Visual Analogic Scale of joint swelling 0-10cm) and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint)) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between joint goniometry(°) and ultrasonography findings ( determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between use of analgesics(tablets per day of paracetamol) and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between handgrip strength determined by Jamar dynamometer grip(kgf) and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between pinch strength determined by the dynamometer of Pinch Gauge(kgf) and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between hand function(determined by AUSCANindex and COCHIN questionnaire) and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks
Change from baseline - Correlation between VAS of the joint on movement and ultrasonography findings(determined using the Grey Scale and power Doppler in affected joint) at 1year in six times | 0,1,4,8,12 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rita NV Furtado, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Rheumatology of Federal University of São Paulo, São Paulo, São Paulo, Brazil